CLINICAL TRIAL: NCT02065466
Title: A Pilot Study of the Combination of Nab-paclitaxel, Temozolomide and Bevacizumab in Patients With Metastatic Melanoma With Brain Metastases
Brief Title: Combo of Abraxane, TMZ, Bevacizumab in Metastatic Melanoma With Brain Metastases
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1312169092
Record Dates: First submitted 2014-02-06; First posted 2014-02-19 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Metastatic Melanoma; Brain Metastases
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Temozolomide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination (Experimental): nab-paclitaxel and temozolomide combined with full dose of bevacizumab
  Interventions: Drug: nab-paclitaxel; Drug: Temozolomide; Drug: Bevacizumab

INTERVENTIONS:
Drug: nab-paclitaxel
Drug: Temozolomide
Drug: Bevacizumab

SUMMARY:
1.1. Primary Objectives

1. To determine if nab-paclitaxel and temozolomide can be combined with full dose of bevacizumab for the therapy of patients with newly diagnosed brain metastases of metastatic malignant melanoma.

* To define the MTD of the combination (Phase I component).
* To determine progression free survival (Phase II component). 1.2. Secondary Objectives

  1. To separately evaluate the response rate and duration of both the brain and extra-cranial systemic metastases.
  2. To define the toxicity of the regimen.
  3. To tabulate the toxicity of the radiotherapy to the brain and compare with known toxicities of radiotherapy to the brain in melanoma and brain metastases.
  4. To use the data generated to plan definitive controlled clinical trials of the combination.
  5. To determine the overall response rate (Phase II component).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed malignant melanoma and clinical evidence of metastatic disease to the brain. Mucosal and ocular melanomas are included.
* Newly developed inoperable brain metastases without associated hemorrhage or midline shift.
* Inoperable or metastatic extra cranial stage III or IV disease.
* Diagnostic quality MRI of the brain or if contraindicated then contrast CT scan of the head performed within 28 days prior to registration.
* Measurable metastases to the brain, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >10 mm in the brain MRI/CT scan.
* CT scan chest, abdomen and pelvis or PET CT scan performed within 28 days of study registration. For disease outside the brain, tumors must be > 10 mm by CT scan.
* Prior therapy allowed but no prior therapy with nab-paclitaxel, paclitaxel, temozolomide, DTIC or bevacizumab.
* Bevacizumab may not be initiated until 4 weeks after surgical resection or radiation therapy completion.
* Age 18 or older.
* Pre-existing peripheral neuropathy must have < Grade 2 (per CTCAE 4.0) at the time of registration.
* Negative serum or urine β-hCG pregnancy test at screening for patients of childbearing potential.
* Women of childbearing potential and sexually active males must use an effective contraception method during treatment and for three months after completing treatment.
* ECOG Performance status 0-1.
* Estimated life expectancy of greater than 2 months.
* Patients must have adequate organ function as defined below (these must be evaluated within 14 days prior to registration):
* leukocytes >3,000/mcL
* absolute neutrophil count >1,500/mcL
* platelets >100,000/mcL
* Hemoglobin >9.0 g/dL
* AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit
* Alkaline phosphatase <2.5 X institutional upper limit
* Total bilirubin <1.5 X institutional upper limit of normal (unless associated with Gilbert's syndrome)
* serum creatinine < 1.5 mg/dL OR 1.5 x institutional normal
* LDH there is no restriction
* INR <1.5 PTT WNL
* Urine protein (UPC) ratio 1.0 OR
* Urine dipstick for proteinuria. Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
* Able to render informed consent.

Exclusion Criteria:

* Prior surgical resection for brain metastases.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab, nab-paclitaxel or temozolomide.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring parenteral antibiotics, symptomatic congestive heart failure, unstable angina pectoris, untreated cardiac arrhythmia and peripheral vascular disease.
* History of myocardial infarction or unstable angina within 6 months prior to Day 1.
* History of stroke or transient ischemic attack within 6 months prior to Day 1.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study screening.
* Serious, non-healed wound, ulcer, or bone fracture.
* History of hepatitis B, C or HIV.
* Uncontrolled hypertension or chronic renal disease. No known bleeding diathesis.
* Known hypersensitivity to human albumin.
* Surgery within 4 weeks of study registration. Must be fully recovered and fully healed from any prior surgery.
* Patients having chemotherapy or extra cranial radiotherapy within 4 weeks prior to study screening or those who have not recovered from adverse events due to agents administered more than 4 weeks prior to the completion of study screening.
* Evidence of other concurrent active malignancy.
* Pregnant or nursing.
* Not be receiving any other investigational agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerance Dose | Beginning of Treatment to unstable disease or discontinuation (6 months)
  To define the MTD of the combination (Phase I component).
Progression Free Survival | Treatment to End of Follow-up (6 Months)
  To determine progression free survival (Phase II component).

SECONDARY OUTCOMES:
Response Rate | Baseline to end of follow-up (six months)
  To determine the overall response rate (Phase II component).

CONTACTS AND LOCATIONS:
Overall Officials: Lee Cranmer, MD, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona